CLINICAL TRIAL: NCT06747468
Title: A Phase 3 Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Avexitide in Participants With Post-Bariatric Hypoglycemia
Brief Title: Avexitide for Treatment of Post-Bariatric Hypoglycemia
Acronym: LUCIDITY
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amylyx Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AVX-001
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Post Bariatric Hypoglycemia
Keywords: avexitide; post bariatric hypoglycemia; PBH; hypoglycemia; hypoglycemia post bariatric surgery; Roux-en-Y gastric bypass (RYGB); RYGB; AVX; LUCIDITY; exendin 9-39; exendin; exendin 939; Roux-en-Y; gastric bypass; low blood sugar; Roux-en-Y gastric bypass
MeSH Terms: conditions — Hypoglycemia | interventions — exendin (9-39)

STUDY DESIGN:
Intervention Model Description: Upon entering the Double-Blind period, approximately 75 participants will be randomized and assigned in a 3:2 ratio to either the avexitide treatment group or the placebo group, respectively.
Who Masked: Participant, Investigator
Masking Description: Sponsor, Participant and Investigator are all masked to treatment assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- AVEXITIDE (Experimental): Avexitide (90 mg via subcutaneous [SC] injection) will be taken once per day, in the morning at least 60 minutes before the morning meal, through the duration of the treatment and OLE periods.
  Interventions: Drug: Avexitide
- PLACEBO (Placebo Comparator): Placebo will be taken once per day, via subcutaneous [SC] injection, in the morning at least 60 minutes before the morning meal, through the duration of the treatment period.
  Participants receiving Placebo in the double-blind treatment period will transition to Avexitide 90 mg (via subcutaneous [SC] injection) in the open-label extension (OLE) period.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Avexitide — Avexitide (also known as exendin 9-39), a first-in-class glucagon-like peptide-1 (GLP-1) receptor antagonist, is a 31-amino acid peptide with a free amino group at the N-terminus and an amidated C-terminus. By binding to the GLP-1 receptor, avexitide inhibits GLP-1 receptor signaling, thereby reducing GLP-1 receptor-mediated insulin secretion
  Other Names: exendin 9-39
  Arms: AVEXITIDE
Other: Placebo — Matching placebo comparator
  Arms: PLACEBO

SUMMARY:
AVX-001 (LUCIDITY) is a Phase 3 study to evaluate avexitide compared to placebo in participants with post bariatric hypoglycemia (PBH) related to Roux-en-Y gastric bypass (RYGB). The study will assess avexitide compared to placebo for safety and efficacy, measured by reduction of hypoglycemic events. The study includes a Screening period with a Run-in period (of up to 6- and 3-weeks, respectively); a randomized, double-blind, placebo-controlled study treatment period of 16 weeks; and a two-part open-label extension (OLE) period with a duration of approximately 32 weeks.

DETAILED DESCRIPTION:
AVX-001 (LUCIDITY) is a Phase 3 multicenter study to evaluate avexitide compared to placebo in participants with post bariatric hypoglycemia (PBH) related to Roux-en-Y gastric bypass (RYGB).

Eligible participants must have a confirmed diagnosis of PBH related to RYGB, must be a minimum of 1-year post-surgery, and must have experienced at least 3 discrete hypoglycemic events during the 3-week study Run-in period while adhering to consistent dietary management.

The study includes a Screening period of up to 6 weeks in duration, inclusive of a 3-week Run-in period; a randomized, double-blind, placebo-controlled study treatment period of 16 weeks in duration; and a two-part open-label extension (OLE) period with a duration of 32 weeks.

The Double-Blind period is designed to evaluate the efficacy and safety of 90 mg per day of avexitide (given by subcutaneous injection) compared to placebo in participants with PBH after Roux-en-Y gastric bypass (RYGB), who are not adequately controlled on dietary management for reduction of hypoglycemic events.

The subsequent 32-week Open Label Extension (OLE) period is intended to further evaluate the safety and efficacy of avexitide (90 mg per day, given by subcutaneous injection) in participants who have completed the Double-Blind period. The OLE period consists of an 8-week initial Part A and a subsequent 24-week Part B.

Participants will use a continuous glucose monitor (CGM) in blinded mode, a self-monitoring of blood glucose (SMBG) device (glucose meter), and an electronic diary (eDiary) on a smartphone to record hypoglycemic events and study drug administration during the screening period, 16-week double-blind period, and 8-week OLE Part A. While the CGM is in blinded mode, participants will not see their specific blood glucose values on their CGM, but they will receive an alert when their blood glucose is low; they may check their blood glucose via the SMBG glucose meter device at any time. During the 24-week OLE Part B, participants will use a CGM in unblinded mode (blood glucose values are visible to the participant) and the SMBG and eDiary devices will not be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent and understand the purpose and risks of the study
* Willing and able to adhere to study requirements, including the use of the study-provided CGM device, SMBG device, and eDiary device as well as the other study evaluations and procedures.
* Is male or female, at least 18 years of age (inclusive) at the time of consent.
* Body mass index (BMI) of up to 40 kg/m2 and has stable body weight-i.e., not varying by >5% for at least 2 months prior to Screening
* Has undergone documented RYGB performed ≥12 months prior to Screening.
* Has clinical diagnosis of PBH-defined as history of recurrent hypoglycemia with onset after surgery and having ruled out other causes of hypoglycemia as per Investigator judgment.
* Has recurrent hypoglycemia, as demonstrated by experiencing at least 3 discrete hypoglycemic episodes during the 3-week study Run-in period.
* Must agree to consistently follow the dietary management guidance and to maintain consistent exercise and/or physical activity level throughout the Screening period (including the Run-in period), the Double-Blind study treatment period, and Part A of the OLE period.
* If female, must meet all of the following:

  * Is not breastfeeding or lactating;
  * If of childbearing potential, has negative serum pregnancy test result at Screening and on Day 1 ahead of dosing
  * If of childbearing potential, must also agree to use a highly effective method of birth control-and agree not to participate in egg (ova) donation or storage, throughout the duration of study participation and for at least 1 month after the last dose of study drug.
* If male and engaging in heterosexual intercourse with a female partner of childbearing potential, must utilize a highly effective method of contraception, and agree not to donate sperm, from the time of providing written informed consent until at least 3 months after the last dose of study drug.

Exclusion Criteria:

* Has received avexitide (exendin 9-39) at any time prior to Screening Visit 1.
* Has received another investigational drug, for any indication, within 5 half-lives of that drug prior to Screening Visit 1.
* Has participated in another interventional clinical study within 30 days prior to Screening Visit 1.
* Presence of gastrostomy tube (G-tube).
* Any known or suspected allergy to one of the investigational medicinal products (avexitide or placebo) or any related product (e.g., exenatide).
* History or presence of insulinoma or other cause of endogenous hyperinsulinism other than PBH.
* Active psychiatric disease or active eating disorder (e.g., uncontrolled major depressive disorder, schizophrenia, bipolar disorder, or other severe mood, anxiety, or eating disorder). Note: prospective participants with stable conditions, per Investigator judgement, may be considered, provided they are not on an excluded medication.
* History of major surgery within 6 months prior to Screening.
* History of upper GI surgery, other than RYGB. Note that history of vertical sleeve gastrectomy (VSG) with subsequent RYGB conversion may be considered on a case-by-case basis upon discussion with the Medical Monitor.
* Current or prior use of agent(s) that may alter glucose metabolism, or promote weight loss, within 5 medication half-lives of Screening Visit 1. Such agents include, but are not limited to, the following: acarbose; calcium channel blockers; diazoxide; dipeptidyl-peptidase-4 (DPP-4) inhibitors; GLP-1 agonists; glucocorticoids; glucose-dependent insulinotropic polypeptide (GIP)/GLP-1 dual agonists; insulin; lithium; meglitinides; metformin; pentamide; sodium-glucose-linked transporter (SGLT)-1 inhibitors; SGLT-2 inhibitors; somatostatin analogs; sulfonylureas; and thiazolidinediones (TZDs).
* Use of drugs that interfere with the Dexcom G7 sensor within 5 half-lives of Screening Visit 1. Such drugs include acetaminophen administered at a dosage greater than 1000 mg every 6 hours, and hydroxyurea.
* Investigator-assessed evidence of alcohol or drug abuse within 12 months prior to Screening. Unwillingness to restrict alcohol use to no more than 1 drink per day is also exclusionary.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Composite rate of Level 2 and Level 3 hypoglycemic events | During the double-blind treatment period (approximately 16 weeks)
  Composite rate of Level 2 hypoglycemia (as measured by self-monitoring of blood glucose [SMBG]) and Level 3 hypoglycemia (per American Diabetes Association [ADA], European Association for the Study of Diabetes [EASD]; adjudicated by independent Event Adjudication Committee [EAC]), assessed during the Double-Blind study treatment period
Safety and Tolerability of avexitide | During the double-blind treatment period (approximately 16 weeks)
  Incidence of adverse events (AEs)-e.g., incidence of treatment-emergent AEs (TEAEs), serious AEs (SAEs), AEs of special interest (AESIs), and TEAEs leading to discontinuation-and other safety assessments (e.g., clinical laboratory results and vital sign measurements), assessed during the Double-Blind study treatment period
Incidence of anti-drug antibodies (ADAb) | During the double-blind treatment period (approximately 16 weeks)
  Incidence of ADAb, assessed during the Double-Blind study treatment period

SECONDARY OUTCOMES:
Further evaluate the efficacy of avexitide compared to placebo for reduction of hypoglycemia | During the double-blind treatment period (approximately 16 weeks)
  Rates of the following, assessed during the Double-Blind study treatment period:
  * Level 2 hypoglycemia as measured by SMBG
  * Level 3 hypoglycemia, adjudicated by EAC
  * Level 2 hypoglycemia as measured by CGM

CONTACTS AND LOCATIONS:
Overall Officials: Amylyx Medical Director, Study Director — Amylyx Pharmaceuticals
Locations (21):
- United States (21):
  - Stanford Health Care - Endocrinology Clinic, Stanford, California
  - University of Colorado Health Anschutz Medical Campus, Aurora, Colorado
  - East Coast Institute for Research, Jacksonville, Florida
  - Hanson Diabetes Center, Port Charlotte, Florida
  - Georgia Clincal Research, Lawrenceville, Georgia
  - Cotton-O'Neil Diabetes and Endocrinology Center, Topeka, Kansas
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts
  - NYC Health + Hospitals/Queens - BRANY, New Hyde Park, New York
  - Duke Center for Metabolic and Weight Loss Surgery, Durham, North Carolina
  - Lucas Research - Morehead City, Morehead City, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Penn Medicine University City, Philadelphia, Pennsylvania
  - Vanderbilt Weight Loss Center, Nashville, Tennessee
  - Endocrine and Psychiatry Center, Houston, Texas
  - Southern Endocrinology & Diabetes Associates, Mesquite, Texas
  - UT Health San Antonio, San Antonio, Texas
  - Diabetes and Gandular Disease Clinic, San Antonio, Texas
  - Consano Clinical Research, Shavano Park, Texas
  - Texas Valley Clinical Research, LLC, Weslaco, Texas
  - UWHealth - Junction Rd Medical Center Endocrinology Clinic, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Proposals for access to IPD by qualified investigators will be reviewed by an independent review committee. Only the de-identified data elements needed to achieve the specific scientific aims of a proposal as outlined in a pre-specified analysis plan will be provided. Study documents such as protocol, SAP, ICF, and CSR, may be provided, if requested and if needed, to conduct the specified analyses.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: TBD: proposals for access to IPD will be reviewed after data is used in regulatory approval in all major countries or regions where filing is planned or after publication, whichever is latest. Exact timing is not currently known.
Access Criteria: Access to IPD will be granted to qualified investigators whose proposed use of the data has been approved by an independent review committee to achieve the aims in their proposal.